CLINICAL TRIAL: NCT06487117
Title: The Efficacy and Safety Assessment of Huafu Shengji Ointment in Patients With Diabetic Foot of Qi Deficiency and Blood Stasis Syndrome: A Study Protocol for a Randomized Controlled Trial
Brief Title: The Efficacy and Safety Assessment of Huafu Shengji Ointment in Patients With Diabetic Foot of Qi Deficiency and Blood Stasis Syndrome
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Daxing District Hospital of Integrated Chinese and Western Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yu Cai, Attending Physician, Beijing Daxing District Hospital of Integrated Chinese and Western Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJB2024030103
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot Ulcer; Huafu Shengji Ointment; Qi Deficiency and Blood Stasis Syndrome; Randomized Controlled Trial
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huafu Shengji Ointment (Experimental): After debridement, Huafu Shengji Ointment is applied topically with a coverage thickness of 1mm, followed by sterile gauze dressing. The dressing is changed every other day. The treatment period is 4-8 weeks.
  Interventions: Drug: Huafu Shengji Ointment
- ethacridine lactate solution (Active Comparator): After debridement, the wound is cleaned and disinfected with ethacridine lactate solution, then covered and dressed with sterile gauze. The dressing is changed every other day. The treatment period is 4-8 weeks.
  Interventions: Drug: ethacridine lactate solution

INTERVENTIONS:
Drug: Huafu Shengji Ointment — Huafu Shengji Ointment
  1. The experimental group received conventional medical treatment: diabetes-related knowledge education, blood sugar control, blood pressure reduction, blood lipid regulation, antiplatelet drugs, vasodilation, nerve nutrition, and the use of antibiotics.
  2. The experimental group receive local debridement: iodophor disinfection, saline cleaning, removal of necrotic tissue, and wound exposure.
  3. After debridement, Huafu Shengji Ointment is applied topically with a coverage thickness of 1mm, followed by sterile gauze dressing. The dressing is changed every other day. The treatment period is 4-8 weeks.
  Arms: Huafu Shengji Ointment
Drug: ethacridine lactate solution — ethacridine lactate solution
  1. The control group received conventional medical treatment: diabetes-related knowledge education, blood sugar control, blood pressure reduction, blood lipid regulation, antiplatelet drugs, vasodilation, nerve nutrition, and the use of antibiotics.
  2. The control group receive local debridement: iodophor disinfection, saline cleaning, removal of necrotic tissue, and wound exposure.
  3. After debridement, the wound is cleaned and disinfected with ethacridine lactate solution, then covered and dressed with sterile gauze. The dressing is changed every other day. The treatment period is 4-8 weeks.
  Arms: ethacridine lactate solution

SUMMARY:
Diabetic foot ulcers, as a complication of diabetes with high disability and mortality rates, have become a significant global healthcare burden and medical challenge worldwide. The clinical situation of chronic non-healing ulcers leading to repeated amputations has not yet been resolved. In preliminary clinical practice, Huafu Shengji Ointment has been shown to significantly improve the complete healing rate of ulcer wounds. This study aims to further comprehensively evaluate the therapeutic effects of Huafu Shengji Ointment and provide high-quality evidence.

ELIGIBILITY:
Inclusion Criteria:

-

Patients who meet the following criteria will be included:

1. Patients who meet the diagnostic criteria for diabetic foot and have a Wagner grade of 1-5.
2. It is in line with the syndrome type of qi deficiency and blood stasis in traditional Chinese medicine.
3. Age between 35 and 80 years
4. The patient had no serious cardiac, liver, renal insufficiency or other systemic infections.
5. No hereditary or infectious diseases, no malignant tumors, and no severe malnutrition in patients.
6. Have understood the treatment modality and voluntarily signed the informed consent form.

Exclusion Criteria:

-

Patients who meet any of the following criteria will be excluded:

1. Patients who experience severe allergic reactions to the experimental medication and cannot undergo treatment.
2. Patients with poorly controlled serious conditions such as diabetic ketoacidosis, ketoacidosis, or diseases of the liver and kidneys.
3. Patients with psychiatric disorders or severe depression.
4. Women who are pregnant or breastfeeding.
5. Patients with severe organic tumors.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ulcer area | Measured once a week, for a total of 8 weeks.
  Method of measuring ulcer area: Sterile transparent dressings are used to trace the edges of the ulcer, digital cameras are used to capture the images, and ImageJ is utilized for analysis and processing.
granulation tissue coverage | Measured once a week, for a total of 8 weeks.
  Granulation tissue area coverage rate = (Area of the wound covered by granulation tissue [mm^2]) / (Total wound area [mm^2]) × 100%
ulcer volume | Measured once a week, for a total of 8 weeks.
  Ulcer volume measurement method: After debridement is completed, the wound surface is dried with a dry cotton ball. Sterile saline is injected into the ulcer cavity using a sterilized syringe until the liquid level is flush with the skin. When the ulcer is a fistula, one end of the fistula is sealed with sterile transparent film, and then saline is injected. The volume of the injected saline is equivalent to the volume of the ulcer.
the time of complete wound healing | complete wound healing (assessed up to 8 weeks)
  Digital cameras capture images, documenting the process of wound from the ulcerative state to the complete in situ healing of the skin tissue.

SECONDARY OUTCOMES:
the skin temperature around the wound | Measured once a week, for a total of 8 weeks.
  0 Normal
  1. Intermittently feels cold
  2. Persistently cold, but can be relieved with warming measures
  3. Persistently cold, and cannot be relieved with warming measures
  4. Even with stronger warming measures than usual in a 20°C environment, still feels cold.
the degree of pain | Measured once a week, for a total of 8 weeks.
  0 No pain
  1. Pain occurs with activity or exertion
  2. Intermittent pain at rest
  3. Persistent pain at rest, but tolerable
  4. Severe persistent pain, sleepless nights, and pain relief requires analgesics
skin color | Measured once a week, for a total of 8 weeks.
  0 Normal skin color
  1. Intermittently pale skin
  2. Persistently pale skin
  3. Skin appears purplish-cyanotic
  4. Skin appears purplish-black or black
the extent of wound exudate | Measured once a week, for a total of 8 weeks.
  Covered with a 10 cm × 10 cm single-layer sterile gauze, scored based on the number of layers of gauze soaked through by exudate over 24 hours 0 1 layer
  1. 2 layers
  2. 3 layers
  3. 4 layers
  4. ≥ 5 layers
alanine aminotransferase | Measured once a week, for a total of 8 weeks.
  The reference range is 0-40 U/L.
aspartate aminotransferase | Measured once a week, for a total of 8 weeks.
  The reference range is 0-40 U/L.
urea nitrogen | Measured once a week, for a total of 8 weeks.
  Reference range value 3.2-7.1 mmol/L
serum creatinine | Measured once a week, for a total of 8 weeks.
  Reference range value: Males 53-106 μmol/L, Females 44-97 μmol/L
electrocardiogram | Measured once a week, for a total of 8 weeks.
  During the study period, the P wave, P-R interval, QRS complex, and QT interval of the electrocardiogram will be assessed.

REFERENCES:
- [Background] Monaghan MG, Borah R, Thomsen C, Browne S. Thou shall not heal: Overcoming the non-healing behaviour of diabetic foot ulcers by engineering the inflammatory microenvironment. Adv Drug Deliv Rev. 2023 Dec;203:115120. doi: 10.1016/j.addr.2023.115120. Epub 2023 Oct 25. PMID 37884128
- [Background] Ibrahim A. IDF Clinical Practice Recommendation on the Diabetic Foot: A guide for healthcare professionals. Diabetes Res Clin Pract. 2017 May;127:285-287. doi: 10.1016/j.diabres.2017.04.013. Epub 2017 Apr 9. No abstract available. PMID 28495183
- [Background] Jupiter DC, Thorud JC, Buckley CJ, Shibuya N. The impact of foot ulceration and amputation on mortality in diabetic patients. I: From ulceration to death, a systematic review. Int Wound J. 2016 Oct;13(5):892-903. doi: 10.1111/iwj.12404. Epub 2015 Jan 20. PMID 25601358
- [Background] Huang YY, Lin CW, Cheng NC, Cazzell SM, Chen HH, Huang KF, Tung KY, Huang HL, Lin PY, Perng CK, Shi B, Liu C, Ma Y, Cao Y, Li Y, Xue Y, Yan L, Li Q, Ning G, Chang SC. Effect of a Novel Macrophage-Regulating Drug on Wound Healing in Patients With Diabetic Foot Ulcers: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2122607. doi: 10.1001/jamanetworkopen.2021.22607. PMID 34477854